CLINICAL TRIAL: NCT02484274
Title: Iron Deficiency in Infants : Population-wide Study of the Protective Role of Toddler Milk Formula
Brief Title: Iron Deficiency (ID) in Infants
Acronym: CARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other); Association Française de Pédiatrie Ambulatoire- AFPA (Unknown); CERBA (Unknown); Laboratoire de Biochimie, CHU Louis Mourier (Unknown); INSERM 1153, Centre de Recherche Epidémiologique et Biostatistique (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P140314
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Iron Deficiency in Young Children Living in France
Keywords: iron-deficiency; iron-deficiency anemia; infants and toddlers; industrialised countries; population-based study; prevalence and risk factors; screening strategies; diagnosis markers; primary prevention
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- infants followed by pediatrician (Other)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — 1 blood sample of 9 ml. 3-day food diary , according to the European Food Safety Authority methodology

SUMMARY:
ID in children is the most frequent micronutrient deficiency in industrialized countries, including France. ID induces neurological impairment reducing cognitive, motor, and behavioral capacities in children in the short and long term.

The purpose of this study is to evaluate the principal determinants of ID in France in two-year-old children and to improve strategies for prevention and screening.

The main objective is to study the association between iron status in two-year-old infants living in France and the consumption of toddler milk formula after taking non-dairy iron ingestion, parental socioeconomic status and educational level into account.

The secondary objectives are the following :

* to estimate the prevalence of ID and ID anemia in 2-year-old children living in France.
* to improve clinical tools for ID screening. to improve strategies for laboratory screening.

DETAILED DESCRIPTION:
The general methodology planned is a nationwide observational cross-sectional study including a blood sample and nutritional survey. 100 pediatricians will include children from 21 regions different from a geographic and a dietary point of view. Each pediatrician will include 10 children consecutively including 3 with the french medical healthcare coverage called CMU (which is a precariousness marker).

The study will take place according to the following plan and procedures for each child: D1 recruitment in the physician-investigator's office (verification of inclusion criteria and collection of the first parent's consent, clinical data collection, prescription for blood test and delivery of the kit containing the elements needed for the study for the patients); between D8 and D15, performance of the standard laboratory tests to be performed locally in the medical laboratory normally used by the family, and the sending of samples for specific analyses (especially biochemistry) to reference laboratory that will perform all these analyses for this study; between D2 and D7, a 3-day food survey based on a food diary (see below); between D20 and D60, final study visit to the doctor's office (help in completing the food diary, discussion of the laboratory results, prescription of iron treatment if needed). The blood sample and/or the 3-days food survey will be delayed 15 days if any intercurrent disease which may interfere with biological markers or food intake (for example acute gastro-enteritis, fever) appears after D1 of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 22-26 months
* living usually in France
* written agreement of one parent or the holder of parental authority
* followed-up by a liberal paediatrician
* with social coverage

Exclusion Criteria:

* chronic disease known at inclusion that might affect iron metabolism or reserves : blood transfusion since birth, celiac disease, chronic inflammatory disease, including of the intestines, cystic fibrosis, other enteropathy, enteral nutrition for more than 15 days in the past 6 months, chronic hemolytic diseases, chronic kidney disease, hemophilia, or chronic bleeding, such as ENT or gastrointestinal, hemochromatosis, any malignant condition, or lead poisoning)
* participation to another study

Ages: 22 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 830 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Serum ferritin level | Between day 8 and day 15 (or plus 15 days)
  Iron deficiency determined by serum ferritin level < 10 µg/l with C Reactive Protein (CRP) < 5 mg/l

SECONDARY OUTCOMES:
Haemoglobin blood level | Between day 8 and day 15 (or plus 15 days)
  Iron-deficiency anemia determined by haemoglobin blood level < 11g/dl in infant with iron deficiency
Dosage of biochemical markers (hepcidin, erythrocytic protoporphyrin) | Between day 8 and day 15 (or plus 15 days)
Iron intake related to toddler milk formula | Between day 2 and day 7 (or plus 15 days)
  Food diary
Parents' economical and educational level | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Martin Chalumeau, MD, PhD, Study Director — INSERM UMR 1153
Locations (1):
- Necker-Enfants Malades hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacri AS, Bocquet A, de Montalembert M, Hercberg S, Gouya L, Blondel B, Ganon A, Hebel P, Vincelet C, Thollot F, Rallo M, Gembara P, Levy C, Chalumeau M. Young children formula consumption and iron deficiency at 24 months in the general population: A national-level study. Clin Nutr. 2021 Jan;40(1):166-173. doi: 10.1016/j.clnu.2020.04.041. Epub 2020 May 7. PMID 32507584
- [Background] Sacri AS, Ferreira D, Khoshnood B, Gouya L, Barros H, Chalumeau M. Stability of serum ferritin measured by immunoturbidimetric assay after storage at -80 degrees C for several years. PLoS One. 2017 Dec 11;12(12):e0188332. doi: 10.1371/journal.pone.0188332. eCollection 2017. PMID 29228047
- [Background] Baker RD, Greer FR; Committee on Nutrition American Academy of Pediatrics. Diagnosis and prevention of iron deficiency and iron-deficiency anemia in infants and young children (0-3 years of age). Pediatrics. 2010 Nov;126(5):1040-50. doi: 10.1542/peds.2010-2576. Epub 2010 Oct 5. PMID 20923825
- [Background] Domellof M, Braegger C, Campoy C, Colomb V, Decsi T, Fewtrell M, Hojsak I, Mihatsch W, Molgaard C, Shamir R, Turck D, van Goudoever J; ESPGHAN Committee on Nutrition. Iron requirements of infants and toddlers. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):119-29. doi: 10.1097/MPG.0000000000000206. PMID 24135983
- [Background] Ghisolfi J, Fantino M, Turck D, de Courcy GP, Vidailhet M. Nutrient intakes of children aged 1-2 years as a function of milk consumption, cows' milk or growing-up milk. Public Health Nutr. 2013 Mar;16(3):524-34. doi: 10.1017/S1368980012002893. Epub 2012 Jul 4. PMID 23098567
- [Derived] Guivarch C, Sacri AS, Levy C, Bocquet A, Lapidus N, Hercberg S, Hebel P, Cheve A, Copin C, Zouari M, Gouya L, de Montalembert M, Cohen JF, Chalumeau M. Clinical Prediction of Iron Deficiency at Age 2 Years: A National Cross-sectional Study in France. J Pediatr. 2021 Aug;235:212-219. doi: 10.1016/j.jpeds.2021.03.072. Epub 2021 Apr 6. PMID 33836187